CLINICAL TRIAL: NCT06496529
Title: ExoDoF: Robotic Exoskeleton for Upper Limb Motor Rehabilitation After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: Agencia Nacional de Investigación y Desarrollo (Other)
Responsible Party: Principal Investigator, Pablo Burgos, Principal Investigator. Ph.D, PT., University of Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FONDEF IDeA 2023 ID23I104
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Stroke
Keywords: stroke recovery; motor recovery; upper extremity recovery
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DoF Group (Experimental): The experimental group with control of the degrees of freedom will receive treatment for 4 weeks using an exoskeleton and also it will be supervised by a physiotherapist.The exoskeleton will restrict the movement of the trunk and upper extremity to leave only the joint free to work in the plane of interest. The training will be selective in an articular plane with biofeedback of movement through videogames and external movement sensors installed in the upper extremity. This movement sensor will allow to interact with the videogames through the movement of the trained movement.
  Interventions: Behavioral: DoF intervention
- Task Group (Active Comparator): The group without control of the degrees of freedom (Task Group) will receive a therapeutic intervention equivalent in dose, but without any restriction of joint movement (without the exoskeleton). Each session will be divided into two parts. In the first part, participants will train with combined planes and in a multi-joint manner with the same video games as DoF Group but with the movement sensor in your hand performing 4 direction movements with the upper limb (horizontal, vertical and diagonals).
  In the second training part, patients will perform functional tasks: raise and lower your hand on the table, cleaning a table, put cream on the non-paretic arm, hold a bottle, put a piece of bread or something similar in your mouth, wash your face, brush your hair, store items in a basket, brush teeth, wrote and serve water in glass.
  Interventions: Behavioral: Task intervention

INTERVENTIONS:
Behavioral: DoF intervention — Training of specific uniarticular and single plane movement of the upper limb through an exoskeleton and videogames that will be supervised by a physiotherapist.
  Arms: DoF Group
Behavioral: Task intervention — Training of multiarticular upper limb movements (vertical, horizontal and diagonal) through videogames and also training of functional task (raise and lower your hand on the table, cleaning a table, put cream on the non-paretic arm, hold a bottle, put a piece of bread or something similar in your mouth, wash your face, brush your hair, store items in a basket, brush teeth, wrote and serve water in glass). This activities will be supervised by a physiotherapist.
  Arms: Task Group

SUMMARY:
Two decades ago, the projection of recovery of the upper extremity (UE) after a stroke had a very poor prognosis worldwide. Nowadays, thanks to medical advances and early rehabilitation, the prognosis for recovery has improved; however, there is still a limit that no therapy has been able to overcome, related to spontaneous recovery as part of the natural evolution of the pathophysiological process, rather than with the contribution of rehabilitation. Additionally, existing therapies show partial effectiveness on the recovery of UE function, but do not avoid the use of compensatory strategies or alternatives to normal movement. Given this situation, there is an active search for new therapeutic approaches. In this clinical trial the investigators propose a rehabilitation paradigm that promotes the recovery of control of specific planes of movement through the selective restriction of degrees of freedom, simplifying control demands. The investigators sought to test the hypothesis that people with stroke in the early subacute stage and who present alterations in the movement of the upper extremity, a rehabilitation protocol that reduces the degrees of freedom of the UE and trunk, enables greater recovery of the movement of the UE and less use of compensatory movements compared to a protocol without DoF control. The general objective is to demonstrate the effect of training with restriction of the degrees of freedom of UE and trunk, mediated by an exoskeleton and videogames, on the control of the UE.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ischemic or hemorrhagic stroke with zero to twelve weeks of evolution.
* Subjects with alterations in active voluntary movement of ES with Fugl Meyer less than or equal to 50 points. Strength of shoulder abduction and finger extension from palpable contraction (1 in Medical Research Council (MRC) scale for muscle strength).

Exclusion Criteria:

* Cognitive impairment that prevents signing the informed consent, following the instructions and understanding the procedures. (MOCA < 18).
* Inability to perform activities sitting for more than 90 minutes or inability to perform activities without severe pain (VAS > 6) or having limited reach ranges.
* Have severe visual impairment that does not allow to carry out the activities associated with the task.
* Previous stroke with neurological sequelae in the upper extremity.
* Present bilateral sensorimotor alterations.
* Damage to the cerebellum/peduncles described in the radiological report or classic signs of cerebellar damage (Upper extremity SARA items of 2 or more)

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in UE-FMA at the end of the training | 3 days post training
  Differences between the Upper Extremity Fugl-Meyer Assessment (UE-FMA) at the beginning of the recruitment and at the end of the training
Change in UE-FMA at 6 months post stroke | 180 days post stroke
  Differences between the Upper Extremity Fugl-Meyer Assessment (UE-FMA) at the beginning of the recruitment and at 6 months post stroke

SECONDARY OUTCOMES:
Change in ARAT at the end of the training | 3 days post training
  Differences between the Action Research Arm Test (ARAT) at the beginning of the recruitment and at the end of the training
Change in ARAT at 6 months post stroke | 180 days post stroke
  Differences between the Action Research Arm Test (ARAT) at the beginning of the recruitment and at 6 months post stroke
Change in iCoh at the end of the training | 3 days post training
  Differences between EEG Ipsi-Contralateral Motor Cortex connectivity (iCoh) at the beginning of the training and at the end of the training
Change in iCoh connectivity at 6 months post stroke | 180 days post stroke
  Differences between EEG Ipsi-Contralateral Motor Cortex connectivity (iCoh) at the beginning of the training and at 6 months post stroke
Change in arm kinematics at the end of the training | 3 days post training
  Differences between arm kinematics (shoulder, elbow, wrist and finger angles during reaching and grasping a glass) at the beginning of the training and at the end of the training
Change in arm kinematics at 6 months post stroke | 180 days post stroke
  Differences between arm kinematics (shoulder, elbow, wrist and finger angles during reaching and grasping a glass) at the beginning of the training and at 6 months post stroke

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Burgos, PhD, Study Director — University of Chile
Locations (4):
- Chile (4):
  - Hospital Clínico Universidad de Chile, Santiago
  - Hospital El Carmen, Santiago
  - Hospital San José, Santiago
  - Hospital Dr. Hernán Henríquez Aravena, Temuco

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After the publication of the clinical trial, for 5 years.
Access Criteria: Based on reasonable request to the project director (Pablo Burgos, pburgos@uchile.cl), the data will be shared.